CLINICAL TRIAL: NCT01783470
Title: Effects of b3-Adrenergic Receptor Agonists on Brown Adipose Tissue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aaron Cypess (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Aaron Cypess, Investigator, NIDDK, NIH, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012P000309; 2P30DK036836-26 (NIH)
Record Dates: First submitted 2013-01-29; First posted 2013-02-05 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Obesity
Keywords: adipose tissue, brown; obesity; Adrenergic beta-3 Receptor Agonists; thermogenesis; metabolism
MeSH Terms: conditions — Obesity | interventions — Adrenergic beta-3 Receptor Agonists; mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- beta3-adrenergic receptor agonist (Experimental): single dose. Each subject was randomized to receive placebo at one visit and then the beta3-adrenergic receptor agonist on another study day.
  Interventions: Drug: beta3-adrenergic receptor agonist

INTERVENTIONS:
Drug: beta3-adrenergic receptor agonist — single dose. The subjects were randomized to receive placebo on one study day and active beta3-adrenergic receptor agonist on the other study day.
  Other Names: mirabegron, which is Myrbetriq (TM) by Astellas Pharma

SUMMARY:
This study will test the hypothesis that human brown adipose tissue (BAT) can be activated using a β3-adrenergic receptor (AR) agonist. The efficacy of β3-AR agonist will be compared with cold exposure, which we have already shown can activate human BAT, as well as a placebo control.

DETAILED DESCRIPTION:
This study will include an outpatient screening visit and three separate, independent overnight study visits in the General Clinical Research Center (GCRC) at Beth Israel Deaconess Medical Center (BIDMC). Screening procedures will consist of a medical history, physical examination, blood draw, and ECG. If, from the screening tests, it is determined that the eligibility criteria have been meet, healthy volunteers will participate in three separate inpatient visits at BIDMC. Study procedures will occur in the GCRC and the Nuclear Medicine suite at BIDMC.

Volunteers will first complete Day A, in which we will measure BAT volume and activity during cold exposure. Cold exposure will consist of wearing a cooling vest at 55 - 61°F, a temperature shown to be cool enough to activate brown adipose tissue but warm enough not to lead to shivering. Resting metabolic rate (RMR) will be measured by indirect calorimetry before and during cool exposure.

If there is detectable brown fat activity on Day A, volunteers will participate in Days B and C. Days B and C will be conducted in random order to reduce any bias from the sequence of treatment and scans, as well as any potential placebo effects. Day B will consist of pharmacological stimulation with β3-AR agonist. On Day C, volunteers will be given a placebo control and will not undergo cooling.

A blood draw of 26 cc will always be done prior to FDG injection and FDG PET/CT will always be performed 60 minutes after FDG injection. On Day A, FDG will be injected after 60 minutes of cool exposure and the volunteer will remain in the cooling vest for another 60 minutes after FDG injection.

To compare energy expenditure and BAT mass and activity among volunteers, we will normalize the data to fat and muscle mass. Whole-body and regional fat and muscle mass will be measured via a Dual Energy X-ray Absorptiometry (DXA) scan at the end of Day A.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male
* 18-65 years old
* BMI between 18-40
* Not participated in clinical trial and received either an investigational or marketed drug within two months prior to the study
* Not donated blood in previous two months

Exclusion Criteria:

* Women
* History of local or systemic infection disease with fever or requiring antibiotic within 4 weeks of drug administration
* Corrected QT interval above normal
* Laboratory test results that is more than 1.5 fold outside normal range and/or is judged to be clinically significant
* Current addition to alcohol or substances of abuse
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Use of system course of corticosteroids or other medication known to cause insulin resistance in previous 6 weeks
* Hyperthyroidism,hypothyroidism, hypertension (even if controlled with medications), heart disease (including CAD and CHF), cardiac arrhythmias, diabetes, unstable vasomotor system, or use of monoamine oxidase (MAO) inhibitors
* Diagnosis of bladder outlet obstruction or use of any medication to treat overactive bladder (e.g. Tolterodine, Solifenacin, Propiverine, Oxybutynin, and Fesoterodine)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron M Cypess, MD PhD, Principal Investigator — NIDDK, NIH
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cypess AM, Weiner LS, Roberts-Toler C, Franquet Elia E, Kessler SH, Kahn PA, English J, Chatman K, Trauger SA, Doria A, Kolodny GM. Activation of human brown adipose tissue by a beta3-adrenergic receptor agonist. Cell Metab. 2015 Jan 6;21(1):33-8. doi: 10.1016/j.cmet.2014.12.009. PMID 25565203

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 15 participants who were enrolled. Three of them did not have cold-induced detectable brown fat, so they did not continue to the randomization. The remaining 12 participants had cold-induced brown fat, so they were randomized.
Groups:
- Placebo Then beta3-adrenergic Receptor (AR) Agonist: Participants administered a lactose-based oral placebo followed by administration of the PET tracer FDG and then PET/CT scanning. On a subsequent day that was at least 48 hours later (for washout purposes) these subjects then received drug.
- beta3-adrenergic Receptor (AR) Agonist Then Placebo: Participants administered an oral beta3-AR agonist followed by administration of the PET tracer FDG and then PET/CT scanning. On a subsequent day that was at least 48 hours later (for washout purposes) these subjects then received placebo.
Period: Overall Study
Arm/Group | Placebo Then beta3-adrenergic Receptor (AR) Agonist | beta3-adrenergic Receptor (AR) Agonist Then Placebo
Started | 6 | 6 (Single-dose)
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants randomized to placebo or drug first then received the other treatment second.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.2 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: BAT Activity as Measured by 18F-FDG PET/CT
Description: difference in BAT metabolic activity measured in placebo and active drug arms. The BAT metabolic activity represents the amount of FDG tracer retained within the tissue. Retained FDG is a biomarker for tissue oxygen consumption and hence energy expenditure by the tissue.
Time Frame: 60 min after FDG administration
Measure: Median (Inter-Quartile Range); unit: mL*SUVmean*g/mL
Groups:
- Placebo: lactose
  Placebo
Arm/Group | Placebo | beta3-adrenergic Receptor (AR)
Number analyzed (Participants) | 12 | 12
mL*SUVmean*g/mL | 0.92 [0.48 to 2.82] | 132 [70 to 253]
Statistical Analysis 1: Comparison: Placebo vs beta3-adrenergic Receptor (AR); Since the sample size of twelve subjects limited the ability to demonstrate that measurements were normally distributed, we used the non-parametric Wilcoxon sign-ranks test to assess the primary and secondary endpoints. All p values presented are two tailed. p values < 0.05 were considered to indicate statistical significance for the primary outcome; Test type: Equivalence — All p values presented are two tailed. p values < 0.05 were considered to indicate statistical significance for the primary outcome; p = 0.001, Wilcoxon sign-ranks test

2. Other Pre Specified Outcome: Whole-body Energy Expenditure
Description: This is the energy expenditure as calculated using indirect calorimetry.
Time Frame: 30 minutes before drug administration followed by 30 minutes after FDG administration
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- beta3-adrenergic Receptor Agonist: single dose
  beta3-adrenergic receptor agonist: single dose
- Mild Cold Exposure: 2 hours while wearing a cooling vest with water set to 14-16 C. This arm was before randomization and had 15 participants.
Arm/Group | Placebo | beta3-adrenergic Receptor Agonist | Mild Cold Exposure
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No